CLINICAL TRIAL: NCT00626158
Title: A Phase I Study, With Expanded Cohort, of Biweekly Fixed-dose Rate Gemcitabine Plus Capecitabine in Patients With Advanced Pancreatic and Biliary Carcinomas
Brief Title: Gemcitabine and Capecitabine to Treat Patients With Advanced Pancreatic and Biliary Cancers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: National Comprehensive Cancer Network (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CC#074510
Record Dates: First submitted 2008-02-14; First posted 2008-02-29 (Estimated); Last update posted 2012-04-04 (Estimated); Status verified 2012-04

CONDITIONS: Pancreatic Cancer; Biliary Cancer
Keywords: pancreatic cancer; biliary cancer; gemcitabine; capecitabine
MeSH Terms: conditions — Pancreatic Neoplasms; Biliary Tract Neoplasms | interventions — Gemcitabine; Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Gem/Cape (Experimental)
  Interventions: Drug: gemcitabine; Drug: capecitabine

INTERVENTIONS:
Drug: gemcitabine — 1000 mg/m2 IV day 1 of every cycle for 100 minutes (each cycle 14 days)
  Other Names: gemzar
Drug: capecitabine — starting dose 1000 mg/m2 PO twice a day for days 1-7 of each cycle (each cycle 14 days)
  Other Names: xeloda

SUMMARY:
The purpose of this study is to find out what effects gemcitabine plus capecitabine has on patients with pancreatic or biliary cancer, and to determine the optimal dose that can be given safely of these two drugs together (called the maximum tolerated dose). Gemcitabine and capecitabine are two chemotherapy drugs used to treat pancreatic and biliary cancer. These two drugs used together are considered an acceptable standard of care for pancreatic and biliary cancers. However, in this study the dose and dosing schedule will be changed, in the hopes that the drugs will have more effect with fewer side effects than when given in the standard way.

ELIGIBILITY:
Inclusion Criteria:

* Histologically-confirmed pancreatic adenocarcinoma or biliary tract carcinoma (cholangiocarcinoma or gallbladder cancer)
* Disease must not be amenable to surgical resection. Patients with either locally advanced or metastatic disease are eligible
* No prior systemic therapy for their diagnosis
* ECOG performance score of 0-1
* Evidence of either or both of the following:

  1. RECIST-defined measurable disease (lesions that can be accurately measured in at least one dimension with the longest diameter ≥ 20mm using conventional techniques or ≥10 mm with spiral CT scan)
  2. An elevated serum CA19-9 at baseline ( ≥ 2X ULN)
* Female patients must be either surgically sterile or postmenopausal, or if of childbearing potential must have a negative pregnancy test (serum or urine) prior to enrollment and agree to use effective barrier contraception during the period of therapy. Oral, implantable, or injectable contraceptives may be affected by cytochrome P450 interactions, and are therefore not considered effective for this study. Male patients must be surgically sterile or must agree to use effective contraception during the period of therapy. The definition of effective contraception will be based on the judgment of the investigator.
* Adequate bone marrow function:

  1. ANC ≥ 1500/uL
  2. platelet count ≥ 100,000/uL
  3. hemoglobin ≥ 9.0 g/dL
* Adequate hepatic function:

  1. Total bilirubin ≤ 1.5 X ULN
  2. AST (SGOT) ≤ 2.5 X ULN
  3. ALT (SGPT) ≤ 2.5 X ULN
* Adequate renal function as determined by either:

  1. Calculated or measured creatinine clearance ≥ 40 mL/min (for calculated creatinine clearance, Cockroft-Gault equation will be used)
  2. Serum creatinine ≤ 1.5 X ULN
* Ability to swallow oral medications
* Ability to understand the nature of this study protocol and give written informed consent
* Willingness and ability to comply with scheduled visits, treatment plans, laboratory tests, and other study procedures.

Exclusion Criteria:

* Any prior systemic or investigational therapy for metastatic or locally advanced pancreatic cancer or biliary cancer. Systemic therapy administered alone or in combination with radiation in the adjuvant setting is permissible as long as it was completed > 6 months prior to the time of study enrollment.
* Inability to comply with study and/or follow-up procedures.
* History of other disease, metabolic dysfunction, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that, in the opinion of the investigator, renders the subject at high risk from treatment complications or might affect the interpretation of the results of the study.
* Presence of central nervous system or brain metastases.
* Pregnancy (positive pregnancy test) or lactation.
* Prior malignancy except for adequately treated basal cell skin cancer, in situ cervical cancer, adequately treated Stage I or II cancer from which the patient is currently in complete remission, or any other form of cancer from which the patient has been disease-free for 5 years.
* Clinically significant cardiac disease (e.g. congestive heart failure, symptomatic coronary artery disease and cardiac arrhythmias not well controlled with medication) or myocardial infarction within the last 12 months.
* Lack of physical integrity of the upper gastrointestinal tract or malabsorption syndrome.
* Known, existing uncontrolled coagulopathy.
* Major surgery within 4 weeks of the start of study treatment, without complete recovery.
* Concurrent/pre-existing use of coumadin.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2008-02; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
To establish the maximum tolerated dose of fixed-dose rate gemcitabine plus capecitabine given by biweekly administration in patients with advanced pancreatic and biliary tract malignancies. | 2 years

SECONDARY OUTCOMES:
Objective response rate (ORR) and disease control rate (DCR) in patients with measurable disease at baseline | 2 years
Biomarker (CA19-9) response rate (decline by ≥ 50%) in patients with elevated CA19-9 (≥ 2x ULN) at baseline. | 2 years
Time to tumor progression (TTP) | 2 years
Overall survival | 2 years
Frequency, type, and grade of adverse events using this combination in this patient population | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Ko, MD, Principal Investigator — University of California, San Francisco
Locations (2):
- United States (2):
  - UCSF Helen Diller Family Comprehensive Cancer Center, San Francisco, California
  - Huntsman Cancer Center, University of Utah, Salt Lake City, Utah